CLINICAL TRIAL: NCT06088706
Title: Evaluation of the Effect of Different Doses of Ozone Therapy on Pain and Function of Patients With Knee Osteoarthritis Referred to the Sports Medicine Clinic of Hazrat Rasool Akram Hospital
Brief Title: Evaluation of the Effect of Different Doses of Ozone Therapy on Pain and Function of Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmad Nazari (Other)
Responsible Party: Sponsor-Investigator, Ahmad Nazari, Assistant Professor, Iran University of Medical Sciences
Organization: Iran University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ir.iums.fmd.rec.1401.412
Record Dates: First submitted 2023-09-28; First posted 2023-10-18 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Intervention Model Description: In the randomized clinical trial study, Convenience Sampling will be done among the patients with knee osteoarthritis called to the sports medicine assessment clinic, at Hazrat Rasool Akram hospital.
  Allocation of patients in treatment groups will be done randomly using blocks with blocks of six in one of the treatment groups as follows:
  A: Control (CL) B: O3 20mg C: O3 40mg
  The block randomization method is used to assign people to the three study groups. For this purpose, the length of the block will be equal to 6 houses (two houses for each treatment).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Clinician: injection interventions are performed under the supervision of a sports medicine specialist who does not know the dose of the injections and only injects the solution prepared by another assistant.
  Assessor Clinician: Assessments before and after interventions will be done by a sports medicine resident who is not involved in running the trial.
  Statistical analyzer: The analysis of the research data will be done by a statistical consultant who is not aware of the patient groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group 1 (O3 20mg) (Experimental): the patient is lying on the bed with his knee flexed at about 45 degrees. Then The syringe containing ozone is prepared by a sports medicine assistant and covered with a label so that the clinician is not aware of the injected ozone dose. Lateral Approach will be used for intra-articular injection. after preparation and drape of the desired position and aspiration, the ozone composition will be injected into the joint. In order to inject for this group, a 10 cc needle and a predetermined concentration of 20 micrograms is injected under sterile conditions. The duration of the injection will be 15-20 seconds. The number of sessions considered for injection will be three sessions, once a week for three weeks. The second and third injection will be done under the same conditions as the first session. In this study, Ozonette Sedecal device ( Spain) will be used. And the exercise therapy protocol is performed.
  Interventions: Procedure: Intra-articular injection of ozone
- Intervention group 2 (O3 40mg) (Active Comparator): Just like intervention group 1, in this group, a predetermined concentration of 40 micrograms ozone is injected under sterile conditions.According to the standard treatment guidelines of the American College of Rheumatology, 1gram of acetaminophen in two doses of 500 mg is allowed up to two weeks after daily injections, which is applicable to all three groups.
  Interventions: Procedure: Intra-articular injection of ozone
- Control group (Placebo Comparator): Just like intervention group 1, in this group, a syringe containing oxygen without ozone is injected under sterile conditions.
  Interventions: Procedure: Intra-articular injection of ozone

INTERVENTIONS:
Procedure: Intra-articular injection of ozone — the patient is lying on the bed with his knee flexed at about 45 degrees. Then The syringe containing ozone is prepared by a sports medicine assistant and covered with a label so that the clinician is not aware of the injected ozone dose. Lateral Approach will be used for intra-articular injection. after preparation and drape of the desired position and aspiration, the ozone composition will be injected into the joint. In order to inject for this group, a 10 cc needle and a predetermined concentration of 20 and 40 micrograms ozone are used under sterile conditions. The duration of the injection will be 15-20 seconds. The number of sessions considered for injection will be three sessions, once a week for three weeks. The second and third injection will be done under the same conditions as the first session. In this study, Ozonette Sedecal device ( Spain) will be used. And the exercise therapy protocol is performed.

SUMMARY:
This study is designed as a randomized clinical trial that will be conducted in Hazrat Rasool Akram Hospital in Tehran. Patients with knee osteoarthritis were selected based on the study entry criteria and written consent was obtained from them. Then, by random assignment, patients will be divided into three treatment groups: control group (under oxygen gas injection), intervention group 1 (intra-articular injection of ozone with a dose of 20 micrograms) and intervention group 2 (intra-articular injection of ozone with a dose of 40 micrograms).

DETAILED DESCRIPTION:
This research is a type of randomized clinical trial (RCT) in which the studied samples will be selected from the patients with knee osteoarthritis referring to Hazrat Rasool Akram hospital by available sampling method. All the stages of this research will be done with the approval of the ethics committee of the Research Vice-Chancellor of Iran University of Medical Sciences, and written consent will be obtained from all the participants in this research.

The population studied in this research will be made up of knee osteoarthritis sufferers who, according to the announcements that will be posted at the hospitals of Iran University of Medical Sciences in Tehran, will come from all urban areas to participate in this study to Hazrat Rasool Akram Hospital.) will be called and after meeting the conditions for entering the research, they will be randomly placed in one of the proposed treatment groups.

The intervention groups in this research are:

1. Control group - intra-articular injection of oxygen without ozone
2. Intervention group 1- Intra-articular injection of ozone with a dose of 20 micrograms
3. Intervention group 2- Intra-articular injection of ozone with a dose of 40 micrograms In the next step, a summary of the evaluation and treatment plans for the participants will be stated in simple language, and after that, the results of the research on the studied patients will be evaluated and the results will be recorded. Then, according to their groups, the patients will be subjected to exercise therapy interventions under supervision in the clinic or based on the Internet for six weeks. Before and in the second week, the first month and the third month after the intervention, patients will be evaluated with VAS, knee range of motion, WOMAC questionnaires and functional tests (6MWT and Timed Up and Go Test).

ELIGIBILITY:
Inclusion Criteria:

* Having primary knee osteoarthritis grade 2 and 3 according to the doctor's diagnosis and based on the Kellgren and Lawrence criteria (the presence of knee pain, morning dryness for less than 30 minutes, crypts during movement and radiological signs of osteoarthritis including joint space reduction, subchondral bone sclerosis and osteophyte formation in knee)
* Age 50-75 years
* Suffering from continuous knee pain for at least six months and with a severity of at least 4 based on the VAS criteria in physical activities such as going up and down the stairs, sitting for a long time and squatting
* Ability to walk independently for at least 30 meters
* Body mass index equal to or less than 35
* Complete consent of the patient to participate in the research
* Balanced mental state

Exclusion Criteria:

* History of intra-articular injections in the knee during the last six months
* Suffering from neuromuscular diseases
* Presence of acute traumatic injury in other ligaments and structures of the knee joint as confirmed by a specialist doctor
* History of previous surgery or injury in the knee and other joints of the lower limbs during the last year
* Presence of bone implants
* The presence of new fractures in the lower limbs during the last year
* Getting malignant tumors
* Participation in sports therapy and physiotherapy programs during the last three months

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Questionnaire evaluations womac | before the intervention and two weeks later, one month and three months after the intervention
  Western Ontario and McMaster Universities Osteoarthritis Index questionnaire or WOMAC for short:
  This questionnaire has 24 items which are arranged in three sections.
  1. The first part examines pain with five items in different positions of walking, climbing stairs, while resting in bed, while sitting or sleeping, and standing.
  2. The second part examines morning dryness and joint stiffness at the end of the day with two items.
  3. The third section examines the patient's functional activities in different situations with seventeen items.
  It is worth mentioning that the translation, localization and validation of WOMAC questionnaire in Iran was done in 2014 by Dr. Ebrahimzadeh and his colleagues.
Visual Analogue Scale | before the intervention and two weeks later, one month and three months after the intervention
  Feeling pain in the knee with vas criteria

SECONDARY OUTCOMES:
range of motion | before the intervention and two weeks later, one month and three months after the intervention
  In this research, the active range of motion of the knee is measured with a goniometer and recorded in degrees
Timed Up & Go functional test | before the intervention and two weeks later, one month and three months after the intervention
  n this evaluation, the patient will be asked to get up from a standard chair and walk along a line drawn on the floor in front of a three-meter long chair in a completely comfortable and safe manner, then go around and walk again. Return to the side of the chair and sit on it. The time to perform this test will be measured with a stopwatch and recorded in seconds.
Six-Minute Walk Functional Test | before the intervention and two weeks later, one month and three months after the intervention
  In this evaluation, the patient will be asked to walk the maximum distance he can within 6 minutes. The distance traveled by the patient during the test will be measured with a tape measure and recorded with a meter unit.
  Each of these functional evaluations is repeated three times and the best result for the patient will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sports and Exercise Medicine, School of Medicine, Iran University of Medical Sciences, Tehran, Iran

REFERENCES:
- [Derived] Arjmanddoust Z, Nazari A, Moezy A. Efficacy of two doses of intra-articular ozone therapy for pain and functional mobility in knee osteoarthritis: a double-blind randomized trial. Adv Rheumatol. 2025 Mar 6;65(1):11. doi: 10.1186/s42358-025-00443-w. PMID 40050950